CLINICAL TRIAL: NCT02097537
Title: Study of Methacholine Chloride Inhalation Challenge in Children With Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MC1002
Record Dates: First submitted 2014-03-19; First posted 2014-03-27 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride

ARMS (1):
- Methacholine Chloride (Experimental): children with bronchial asthma
  Interventions: Drug: Methacholine Chloride (SK-1211)

INTERVENTIONS:
Drug: Methacholine Chloride (SK-1211)

SUMMARY:
The Purpose of this study is to evaluate the safety and efficacy of SK-1211 inhalation challenge in children with bronchial asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchial asthma
* FEV1/FVC must be 70% or more
* <10% decrease in FEV1 in response to inhalation of normal saline

Exclusion Criteria:

* Moderate or severe airflow limitation（FEV1<60% predicted）
* Heart attack or stroke in last 3 months
* Uncontrolled hypertension, systolic BP>200, or diastolic BP>100
* known aortic aneurysm

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Methacholine Chloride: children with bronchial asthma
  Methacholine Chloride (SK-1211)
Period: Overall Study
Arm/Group | Methacholine Chloride
Started (Informed consent) | 10
Enrollment | 10 (Inhalation of Methacholine Chloride)
Follow-Up | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects who have inhaled the investigational drug at least once.
Arm/Group | Methacholine Chloride
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Japan | 10

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Number of Subjects Whose PC20 is Less Than 8 mg/mL
Description: The methacholine challenge test is for assessment of bronchial sensitivity, it is assessed by FEV1 (Forced Expiratory Volume in one second) with spirometer.
  For measurement of FEV1, a patient is inhaled saline as baseline and each dose of methacholine which be gradually diluted, inhalations are discontinued with a drop in FEV1 of 20% or more.
  The concentration of methacholine causing 20% fall in FEV1 is PC20.
Time Frame: Visit 1 (Day 1)
Measure: Number; unit: percentage of the subjects
Arm/Group | Methacholine Chloride
Number analyzed (Participants) | 10
percentage of the subjects | 7

2. Secondary Outcome: The Rate of Subjects Whose FEV1 Falls More Than 20% From Baseline Before the Highest Concentration Inhalation
Time Frame: Visit 1 (Day 1)
Measure: Number; unit: percentage of the subjects
Arm/Group | Methacholine Chloride
Number analyzed (Participants) | 10
percentage of the subjects | 7

3. Secondary Outcome: The Summary Statistics of PC20
Description: PC20 : the concentration of methacholine causing 20% fall in FEV1.
Time Frame: Visit 1 (Day 1)
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Methacholine Chloride
Number analyzed (Participants) | 10
mg/mL | 8.0674 (11.7127)

ADVERSE EVENTS:
Time Frame: Visit 1 (Day 1)
Arm/Group | Methacholine Chloride
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methacholine Chloride (N=10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Breath sounds abnormal (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No